CLINICAL TRIAL: NCT00689052
Title: A Randomized, Double-blind, Placebo-controlled, Dose Titration Efficacy and Safety Study of Pramipexole ER (0.75 to 4.5 mg) Administered Orally Once Daily Versus Placebo Over a 16-week Maintenance Phase in Patients Diagnosed With Fibromyalgia, as Assessed by the American College of Rheumatology (ACR) Criteria Followed by a 24-week Open-label Extension Phase
Brief Title: Pramipexole ER vs. Placebo in Fibromyalgia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 248.637
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2009-11-25 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pramipexole ER (Experimental): 0.75 mg to 4.5 mg tablets of Pramipexole ER, once daily in the evening
  Interventions: Drug: pramipexole ER
- Placebo (Placebo Comparator): Placebo tablets, once daily in the evening
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pramipexole ER
  Arms: Pramipexole ER
Drug: placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the efficacy and safety of an extended-release (ER) formulation of pramipexole in comparison with placebo for the treatment of fibromyalgia.

The objective of the open-label phase is to assess the safety profile and effect of Pramipexole (PPX) extended-release (ER) in fibromyalgia patients over a 24-week period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients greater than or equal to 18 years of age
2. Meet criteria for primary fibromyalgia as defined by the American College of Rheumatology (ACR): widespread aching pain in all four quadrants of the body and axial skeleton for greater than 3 months duration and greater than or equal to 11 of 18 tender points under digital palpitation examination with an approximate force of 4 kilograms per centimeters squared (kg/cm2)
3. Pain score of greater than or equal to 4 (scored once at screening and as a weekly mean at baseline) on the 11-point Likert pain scale with 0 = no pain and 10 = worst possible pain
4. Score of greater than or equal to 4 (= moderately ill) on the Clinical Global Impression of Severity (CGI-S) at screening and at baseline
5. All females of child-bearing potential must test negative for pregnancy at Visit 1. Females of child-bearing potential (not surgically sterilized and between menarche and two years postmenopausal) must agree to utilize medically acceptable and reliable means of birth control as determined by the investigator during the study and for one month following the last dose of study medication. Examples of reliable methods include: use of hormonal contraception (oral, injectable, or subcutaneous), double-barrier method, abstinence, partner with vasectomy, or hormonal intrauterine devices
6. Educational level and degree of understanding such that the patient can communicate intelligibly with the investigator and study coordinator
7. Judged to be reliable and agree to keep all appointments for clinic visits, tests, and procedures required by the protocol

Exclusion Criteria:

1. Employees of Boehringer Ingelheim (BI) (that is, employees, temporary contract workers, or designees responsible for the conduct of the study)
2. Have received treatment within 30 days prior to screening with a drug that has not received regulatory approval for any indication
3. Have previously completed or withdrawn from this study or any other study investigating pramipexole.
4. Any current or previous diagnosis of psychosis, bipolar disorder, or schizoaffective disorder as assessed by the Mini International Neuropsychiatric Interview (MINI)
5. Have any primary anxiety disorder within the past year as assessed by the Mini International Neuropsychiatric Interview (MINI)
6. Have any Diagnosis of Statistical Manual of Mental Diseases, 4th Edition (DSM-IV) Axis II disorder that would interfere with protocol compliance
7. Medium or high risk of suicidality as assessed by the Mini International Neuropsychiatric Interview (MINI)
8. History of substance abuse/dependence within the past year, excluding nicotine and caffeine
9. A positive urine drug screen for any substance of abuse or excluded medication
10. Women who are pregnant or breast-feeding
11. Have pain symptoms related to traumatic injury that will interfere with the interpretation of outcome measures
12. Patients with regional pain syndromes, multiple surgeries or failed back surgery syndrome
13. A confirmed or previous diagnosis of rheumatoid arthritis, inflammatory arthritis, or infectious arthritis, or an autoimmune disease
14. Abnormal C-Reactive Protein, Anti-Nuclear Antibody (ANA), Rheumatoid factor, or Thyroid Stimulating Hormone (TSH)
15. Any serious or unstable medical or psychiatric condition or clinically significant abnormalities in labs at screening that would lead to hospitalization during the course of the study or otherwise compromise study participation
16. Have uncontrolled seizures
17. Taking any prohibited medications that cannot be discontinued at screening
18. Patients who are treatment-refractory or whose response may be compromised by disability compensation issues
19. Patients with frequent or severe allergic reactions to multiple medications
20. Prior or current treatment with pramipexole
21. Clinically significant renal disease
22. Current or previous diagnosis of malignant melanoma
23. Clinically relevant ophthalmopathy
24. Documented sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (42):
- United States (42):
  - 248.637.01009 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 248.637.01033 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 248.637.01045 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 248.637.01034 Boehringer Ingelheim Investigational Site, Hot Springs, Arkansas
  - 248.637.01032 Boehringer Ingelheim Investigational Site, Arcadia, California
  - 248.637.01044 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 248.637.01036 Boehringer Ingelheim Investigational Site, Santa Ana, California
  - 248.637.01042 Boehringer Ingelheim Investigational Site, Englewood, Colorado
  - 248.637.01031 Boehringer Ingelheim Investigational Site, Danbury, Connecticut
  - 248.637.01035 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 248.637.01023 Boehringer Ingelheim Investigational Site, Fort Myers, Florida
  - 248.637.01047 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 248.637.01043 Boehringer Ingelheim Investigational Site, Palm Beach Gardens, Florida
  - 248.637.01040 Boehringer Ingelheim Investigational Site, Sunrise, Florida
  - 248.637.01027 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 248.637.01007 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 248.637.01028 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 248.637.01010 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 248.637.01016 Boehringer Ingelheim Investigational Site, Newton, Massachusetts
  - 248.637.01014 Boehringer Ingelheim Investigational Site, Lansing, Michigan
  - 248.637.01020 Boehringer Ingelheim Investigational Site, Flowood, Mississippi
  - 248.637.01018 Boehringer Ingelheim Investigational Site, Picayune, Mississippi
  - 248.637.01012 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 248.637.01017 Boehringer Ingelheim Investigational Site, Billings, Montana
  - 248.637.01024 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 248.637.01008 Boehringer Ingelheim Investigational Site, Albany, New York
  - 248.637.01002 Boehringer Ingelheim Investigational Site, New York, New York
  - 248.637.01025 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 248.637.01026 Boehringer Ingelheim Investigational Site, Fargo, North Dakota
  - 248.637.01004 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 248.637.01038 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 248.637.01003 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 248.637.01046 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 248.637.01006 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 248.637.01039 Boehringer Ingelheim Investigational Site, Duncansville, Pennsylvania
  - 248.637.01015 Boehringer Ingelheim Investigational Site, Warwick, Rhode Island
  - 248.637.01019 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 248.637.01037 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 248.637.01041 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 248.637.01021 Boehringer Ingelheim Investigational Site, Renton, Washington
  - 248.637.01029 Boehringer Ingelheim Investigational Site, Seattle, Washington
  - 248.637.01011 Boehringer Ingelheim Investigational Site, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients receive placebo in dose up-titration steps
- Pramipexole: Patients receive pramipexole in dose up-titration steps
Period: Overall Study
Arm/Group | Placebo | Pramipexole
Started | 31 | 30
Completed | 0 | 0
Not Completed | 31 | 30
Not completed — Adverse Event | 4 | 6
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Early termination of the trial | 22 | 24

BASELINE CHARACTERISTICS:
Population: Treated Set, All patients randomized and received treatment
Groups:
- Placebo: Patients receiving matching placebo
- Pramipexole: Patients receiving pramipexole
- Total: Total of all reporting groups
Arm/Group | Placebo | Pramipexole | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (10.3) | 50.7 (9.7) | 51.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Change in the Weekly Mean of the 24-hour Average Pain Score From a Daily Diary as Measured by the 11-point Likert Pain Scale
Description: The 11-point Likert Pain Scale is a numerical rating scale completed by the patient that measures the intensity of pain. The intensity scores range from 0 (no pain) to 10 (worst possible pain)
Time Frame: Baseline and Week 29
Population: FAS (All randomized and treated patients with a baseline and at least one post-baseline will be included in the Full Analysis Set (FAS))
Groups:
- Pramipexole: 0.75 mg to 4.5 mg tablets of Pramipexole ER, once daily in the evening
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Proportion of Patients "Very Much Improved" or "Much Improved" on the Patient's Global Impression of Improvement (PGI-I) 7-point Scale
Description: PGI-I is a self-reported scale completed by the patient that measures the degree of improvement at the time of assessment.
  The score ranges from 1 = very much improved to 7 = very much worse
Time Frame: Week 29 (at the end of the maintenance phase)
Population: as for outcome 1
Arm/Group | Pramipexole ER | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: The Short Form 36 (SF-36) Health Survey, Physical Functioning Subscale (Change From Baseline).
Description: The SF-36 Health Survey is a self-administered 36-item instrument completed by the patient .
  SF 36 has subscales as follows: i) physical functioning (PF), ii) role limitations due to physical problems (RP), iii) bodily pain (BP), iv) general health perceptions (GH), v) vitality (VT), vi) social function (SF), vii) role limitations due to emotional problems (RE), viii) mental health (MH),ix)physical component summary (PCS)and x)mental component summary(MCS).
  Among the subscales, Physical functioning was key secondary endpoint while other were additional secondary endpoints.
  Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale, with higher scores indicating better health status or functioning. The number of items per domain varies from 2 to 1
Time Frame: Baseline and Week 29
Population: as for outcome 1
Arm/Group | Pramipexole ER | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: The Proportion of Patients With at Least a 30% or at Least a 50% Improvement Relative to Baseline in Pain (Assessed on the 11-point Likert Pain Scale
Description: 11-Point Likert Pain Scale is a numerical rating scale completed by the patient that measures the intensity of pain. The intensity scores range from: 0 = no pain to 10 = worst possible pain .
Time Frame: Baseline and Week 29
Population: as for outcome 1
Arm/Group | Pramipexole ER | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Fibromyalgia Impact Questionnaire (FIQ) Total Score (Change From Baseline)
Description: FIQ is a self-reported scale completed by the patient that measures patient status, progress, and outcomes over the past week.
  The FIQ is composed of a total of 20 items; the first 11 items measure physical functioning, and each item is rated on a four-point Likert scale. Items 12 and 13 measure the number of days the patient felt well and the number of days the patient felt unable to work due to their fibromyalgia symptoms. Items 14 through 20 are numerical, 11-point Likert scales (marked in 10-point increments) on which the patient rates work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety, and depression. The total score ranges from 0 to 80. A higher score indicates a more negative impact
Time Frame: Baseline and Week 29
Population: as for outcome 1
Arm/Group | Pramipexole ER | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) (Change From Baseline).
Description: The Hospital Anxiety and Depression Scale (HADS) measures the severity of anxiety and depression. The severity score ranges from: 0 = least severe to 3 = most severe. The total score ranges from 0 to 21; the higher the score, the more severe the anxious/depressive symptoms
Time Frame: Baseline and Week 29
Population: as for outcome 1
Arm/Group | Pramipexole ER | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: The Short Form 36 (SF-36) Health Survey (Change From Baseline) (Excluding the Physical Functioning Subscale(PF)).
Description: as for outcome 3
Time Frame: Baseline and Week 29
Population: as for outcome 1
Arm/Group | Pramipexole ER | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Euroqol- 5 Dimensions (EQ-5D) Survey (Change From Baseline)
Description: The Euroqol- 5 Dimension (EQ-5D) Health Survey is a generic, multidimensional, health related, quality-of-life instrument that contains two parts-a health status profile and a visual analog scale (VAS) to rate global health-related quality of life. The profile contains five items corresponding to five health domains- mobility, self-care, usual activities, pain/discomfort, and mood. A single score is generated for each health state. Data from the EQ-5D can be converted into 243 unique health states. For each health state, there exists a corresponding valuation that allows the patient's health to be represented as an index, which is a value between -0.594 and 1; the higher the score, the better the quality of life.
Time Frame: Baseline and Week 29
Population: as for outcome 1
Arm/Group | Pramipexole ER | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Multidimensional Assessment of Fatigue (MAF) Index (Change From Baseline)
Description: The Multidimensional Assessment of Fatigue (MAF) Index is a 16-item, self-reporting instrument designed to collect data on four dimensions of fatigue- severity, distress, degree of interference in activities of daily living, and timing .
Time Frame: Baseline and Week 29
Population: as for outcome 1
Arm/Group | Pramipexole ER | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Medical Outcomes Study (MOS) Sleep Scale (Change From Baseline)
Description: The Medical Outcomes Study (MOS) sleep scale is a 12-item (MOS1 to MOS12) self reporting sleep measure.
Time Frame: Baseline and Week 29
Population: as for outcome 1
Arm/Group | Pramipexole ER | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Clinical Global Impression of Severity (CGI-S Scores)
Description: Clinical Global Impression of Severity (CGI-S) Scale is a clinician's assessment of patient's severity of illness. The score ranges from 1 = normal, not at all ill to 7 = among the most extremely ill patients
Time Frame: Baseline and Week 29
Population: as for outcome 1
Arm/Group | Pramipexole ER | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Frequency of Rescue Medication for Pain
Description: Acetaminophen/paracetamol (maximum of 4 g/day) to be allowed as rescue medication for pain.
Time Frame: Week 29
Population: as for outcome 1
Arm/Group | Pramipexole ER | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in Mean Tender Point Threshold
Description: The Tender Point Pain Threshold will be assessed for all 18 tender points by a study clinician. A dolorimeter will be used to exert the pressure at each point and to measure the threshold reading; when the patient first indicates pain, the threshold will be recorded in kg/sq.cm ;If the patient reports pain before 1.0 kg/sq.cm is reached (>0 kg/sq.cm), 1.0 kg/sq.cm will be entered. If the patient does not report pain when the maximum pressure is applied (10.0 kg/sq.cm),0 (no pain) will be entered.
Time Frame: Baseline and Week 29
Population: as for outcome 1
Arm/Group | Pramipexole ER | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 72 days
Arm/Group | Placebo | Pramipexole
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/30
Other Adverse Events (participants affected / at risk) | 10/31 | 18/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | Pramipexole (N=30)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | Pramipexole (N=30)
insomnia (Psychiatric disorders) | 3 | 5
sleep attacks (Psychiatric disorders) | 0 | 3
somnolence (Nervous system disorders) | 1 | 5
dizziness (Nervous system disorders) | 1 | 2
headache (Nervous system disorders) | 2 | 2
nausea (Gastrointestinal disorders) | 3 | 7
dry mouth (Gastrointestinal disorders) | 0 | 3
Gastrooesophageal disease (Gastrointestinal disorders) | 0 | 2
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
rash (Skin and subcutaneous tissue disorders) | 2 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
fatigue (General disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
Early termination leading to no number of subjects analysed for any outcome measure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.